CLINICAL TRIAL: NCT03206294
Title: Presence of a Clinical Pharmacist in a Cardiology Department: What Impact on the Management of Diabetic Patients Within Care Pathways? Example of Inpatient Cardiac Patients at GHPSJ
Brief Title: Impact of Pharmacist in Cardiology Service
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: PhCardiab
Record Dates: First submitted 2017-06-29; First posted 2017-07-02 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2018-08

CONDITIONS: Cardiomyopathy, Diabetic
MeSH Terms: conditions — Diabetic Cardiomyopathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pharmacist assessment intervention group (Other): St Joseph Hospital pharmacist assess every diabetic patient hospitalized in cardiology service in term of antidiabetic treatment during the hospitalization
  Interventions: Other: pharmacist assessment

INTERVENTIONS:
Other: pharmacist assessment — St Joseph Hospital pharmacist assess every diabetic patient hospitalized in cardiology service in term of antidiabetic treatment during the hospitalization

SUMMARY:
The coverage of the diabetes is a multidisciplinary care, with practitioners' implication(hospital and liberal), and other medical and paramedical profession: doctor, pharmacist, male nurse, nutritionist, etc. In fact there is a real importance of link between hospital and general medecine outside. That's why the pharmacist's presence during the hospitalization seems to be a good alternative to make the link between hospital and the outside pharmacist where patient take his treatment.

Hospital pharmacis proceed to a treatment conciliation at the entrance and at discharge.

By this conciliation the aim of the study is to show and quantify the impact of pharmacist presence on therapeutic target .

ELIGIBILITY:
Inclusion Criteria:

* Diabetes type 2 patient hospitalized in cardiology service
* Hospitalization more than 24 hours
* with insuline or/and oral anti diabetic

Exclusion Criteria:

* diabètes type 1
* iatrogenic hyperglycaemia
* hospitalization for cardia angiography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2017-04-28 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Measurement of biological test glycosylated haemoglobin evolution between the entrance and discharge | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Romain CADOR, MD, Principal Investigator — GHPSJ
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No